CLINICAL TRIAL: NCT03856593
Title: Comparative Effectiveness of Two Letters to Encourage Judicious Prescribing of Opioids: A County-wide Project in Los Angeles
Brief Title: Encouraging Judicious Prescribing of Opioids in Los Angeles County
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UP-19-00172; P30AG024968 (NIH)
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance-Related Disorders
Keywords: Opioids; Safe prescribing
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard letter (Experimental): Prescribers randomized to this arm will be sent the standard letter.
  Interventions: Behavioral: Standard letter
- Comparator letter (Experimental): Prescribers randomized to this arm will be sent the comparator letter.
  Interventions: Behavioral: Comparator letter

INTERVENTIONS:
Behavioral: Standard letter — The standard letter will be signed by the Chief Medical Examiner-Coroner and County Health Officer of Los Angeles County to notify prescribers of the death in their practice. The letter includes the decedent's name, date of birth and date of death, and outlines the annual number and types of prescription drug deaths seen by the medical examiner, discusses the value of and way to access the State's prescription drug monitoring program and includes five Centers for Disease Control and Prevention (CDC) guideline-recommended safe prescribing strategies: 1) Avoid co-prescribing of opioids with benzodiazepines, 2) prescribe minimal dose necessary for acute pain, 3) consider slow tapers with pauses to below 50 morphine milligram equivalents (MME) per day, 4) avoid prescriptions lasting greater than 3-months for pain, and 5) prescribe naloxone in conjunction with opioids for patients taking > 50 MME per day. The letter also states that CURES review is required by law as of October 2, 2018.
  Arms: Standard letter
Behavioral: Comparator letter — The comparator letter includes all the details in the standard letter plus additional text involving an "if/when/then statement" along with an injunction to providers to share safety information with patients so that they identify as a "safe prescriber." Specifically, the additional text reads as follows: When your next patient presents with pain, keep the above 5 recommendations close at hand to assist with their safe care. Also, be comfortable voicing your concern about prescribing safety with them so that they are also aware of the dangers scheduled drugs may carry. "If/when/then" is a form of "pre-suasion" that provides simple rules that tie goals to specific actions and has been used successfully to encourage behavior in many areas including medication adherence and drug abuse rehabilitation.
  Arms: Comparator letter

SUMMARY:
In collaboration with the Los Angeles County Medical Examiner's Office and the State of California's controlled Substance Utilization Review and Evaluation System (CURES), the investigators propose to review opioid poisonings over 12 months and send letters to prescribers in California when at least one of the provider's prescription(s) was filled by a patient who died of an opioid poisoning in Los Angeles County. The letters will be non-judgmental and factual, explaining that a patient of the provider who was being treated with prescription narcotics died of an opioid poisoning. The letters will also encourage judicious prescribing including use of the CURES system before prescribing. The investigators will evaluate physician prescribing practices over 24 months (12 months pre- and 12 months post-letter) using data from the CURES database. The investigators' hypothesis is that letters will make the risk of opioids more cognitively available and that physicians will respond by prescribing opioids more carefully, resulting in fewer deaths due to misuse and more frequent use of the CURES system.

ELIGIBILITY:
The investigators will not be enrolling subjects. This is an evaluation of a public health intervention involving sending prescriber's factual and nonjudgmental letters, signed by the County Medical Examiner, that would state that a patient the provider had treated with controlled substances died of an opioid poisoning.

Inclusion Criteria:

* Prescribers in California for whom at least one of their prescription(s) was filled by a patient who died of an opioid poisoning in Los Angeles County

Exclusion Criteria:

* Prescriber is licensed outside the State of California and does not hold a California license, but the prescription was filled in California
* The prescriber does not have a CURES report on record
* The prescriber has issued only one opioid prescription in the last 12 months since the time of the deceased death (and the prescription was to the deceased)
* Prescriptions with unknown Drug Enforcement Agency (DEA) number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County Medical Examiner's Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doctor JN, Kelley MA, Goldstein NJ, Lucas J, Knight T, Stewart EP. A randomized trial looking at planning prompts to reduce opioid prescribing. Nat Commun. 2024 Jan 12;15(1):263. doi: 10.1038/s41467-023-44573-5. PMID 38216566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Los Angeles Medical Examiner identified 316 decedents from a schedule II-IV Rx overdose from October 2018 to May 2020. 236 received a schedule II-IV Rx in the 12 months prior to their death from 541 prescribers who were randomized to either the standard letter or comparator. 510 of these clinicians prescribed at least one opioid to 219 decedents and were included in the primary analysis. The secondary analysis included 528 clinicians who prescribed a benzodiazepine to 220 decedents.
Groups:
- Standard Letter: The intervention arm will involve letter A sent to prescribers in Los Angeles County.
  Standard Letter: The letter will be signed by the Chief Medical Examiner-Coroner and County Health Officer of Los Angeles County to notify prescribers of the death in their practice. The letter includes the decedent's name, date of birth and date of death, and outlines the annual number and types of prescription drug deaths seen by the medical examiner, discusses the value of and way to access the State's prescription drug monitoring program and includes five Centers for Disease Control and Prevention (CDC) guideline-recommended safe prescribing strategies: 1) Avoid co-prescribing of opioids with benzodiazepines, 2) prescribe minimal dose necessary for acute pain, 3) consider slow tapers with pauses to below 50 MME per day, 4) avoid prescriptions lasting greater than 3-months for pain, and 5) prescribe naloxone in conjunction with opioids for patients taking > 50 MME per day. The letter also states that CURES review is required by law as of October 2, 2018.
- Comparator Letter: The intervention arm will involve the comparator letter B to prescribers in Los Angeles County.
  Comparator Letter: This letter includes all the details in Standard Letter plus additional text involving an "if/when/then statement" along with an injunction to providers to share safety information with patients so that they identify as a "safe prescriber." Specifically, the additional text reads as follows: When your next patient presents with pain, keep the above 5 recommendations close at hand to assist with their safe care. Also, be comfortable voicing your concern about prescribing safety with them so that they are also aware of the dangers scheduled drugs may carry. "If/when/then" is a form of "pre-suasion" that provides simple rules that tie goals to specific actions and has been used successfully to encourage behavior in many areas including medication adherence and drug abuse rehabilitation.
Period: Overall Study
Arm/Group | Standard Letter | Comparator Letter
Started | 284 | 257
Completed | 269 | 241
Not Completed | 15 | 16
Not completed — Prescriber had no opioid prescriptions or was missing prescription information during study period | 15 | 16

BASELINE CHARACTERISTICS:
Groups:
- Standard Letter: The intervention arm will involve the Standard Letter sent to prescribers in Los Angeles County.
  Standard Letter: The letter will be signed by the Chief Medical Examiner-Coroner and County Health Officer of Los Angeles County to notify prescribers of the death in their practice. The letter includes the decedent's name, date of birth and date of death, and outlines the annual number and types of prescription drug deaths seen by the medical examiner, discusses the value of and way to access the State's prescription drug monitoring program and includes five Centers for Disease Control and Prevention (CDC) guideline-recommended safe prescribing strategies: 1) Avoid co-prescribing of opioids with benzodiazepines, 2) prescribe minimal dose necessary for acute pain, 3) consider slow tapers with pauses to below 50 MME per day, 4) avoid prescriptions lasting greater than 3-months for pain, and 5) prescribe naloxone in conjunction with opioids for patients taking > 50 MME per day. The letter also states that CURES review is required by law as of October 2, 2018.
- Comparator Letter: The intervention arm will involve the Comparator Letter sent to prescribers in Los Angeles County.
  Comparator Letter: This letter includes all the details in the Standard Letter plus additional text involving an "if/when/then statement" along with an injunction to providers to share safety information with patients so that they identify as a "safe prescriber." Specifically, the additional text reads as follows: When your next patient presents with pain, keep the above 5 recommendations close at hand to assist with their safe care. Also, be comfortable voicing your concern about prescribing safety with them so that they are also aware of the dangers scheduled drugs may carry. "If/when/then" is a form of "pre-suasion" that provides simple rules that tie goals to specific actions and has been used successfully to encourage behavior in many areas including medication adherence and drug abuse rehabilitation.
- Total: Total of all reporting groups
Arm/Group | Standard Letter | Comparator Letter | Total
Number analyzed (Participants) | 284 | 257 | 541
Age, Categorical [Count of Participants; unit: Participants] — Population: No age data were collected
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some participants are missing biological sex information or declined to disclose.
  Participants
    number analyzed (Participants) | 133 | 126 | 259
    Female | 29 | 27 | 56
    Male | 104 | 99 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 2 | 12
  White | 31 | 22 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 229 | 218 | 447
Region of Enrollment [Number; unit: participants]
  United States | 284 | 257 | 541

OUTCOME MEASURES:

1. Primary Outcome: Average Weekly Change in Morphine Milligram Equivalents (MME) Dispensed
Description: Difference in average weekly MME dispensed 52 weeks pre-letter to 4-52 (excludes 0-3 weeks for washout) post-letter. Measure of interest is the difference in the above measure between prescribers randomized to the standard letter and the comparator letter, referred to as the difference-in-difference (interaction coefficient).
Time Frame: 52 weeks pre-letter to 4-52 weeks post-letter (excludes 0-3 weeks for washout)
Population: Prescribers practicing in Los Angeles County with scheduled drug prescribing privileges who prescribed an opioid 52 weeks (1 year) prior to a patient death from a schedule II-IV overdose.
Measure: Mean (95% Confidence Interval); unit: Estimated average weekly MME dispensed
Groups:
- Standard Letter: This arm will involve the Standard Letter sent to prescribers in Los Angeles County.
  Standard Letter: The letter will be signed by the Chief Medical Examiner-Coroner and County Health Officer of Los Angeles County to notify prescribers of the death in their practice. The letter includes the decedent's name, date of birth and date of death, and outlines the annual number and types of prescription drug deaths seen by the medical examiner, discusses the value of and way to access the State's prescription drug monitoring program and includes five Centers for Disease Control and Prevention (CDC) guideline-recommended safe prescribing strategies: 1) Avoid co-prescribing of opioids with benzodiazepines, 2) prescribe minimal dose necessary for acute pain, 3) consider slow tapers with pauses to below 50 MME per day, 4) avoid prescriptions lasting greater than 3-months for pain, and 5) prescribe naloxone in conjunction with opioids for patients taking > 50 MME per day. The letter also states that CURES review is required by law as of October 2, 2018.
- Comparator Letter: This intervention arm will involve Comparator Letter sent to prescribers in Los Angeles County.
  Comparator Letter: This letter includes all the details in the Standard Letter plus additional text involving an "if/when/then statement" along with an injunction to providers to share safety information with patients so that they identify as a "safe prescriber." Specifically, the additional text reads as follows: When your next patient presents with pain, keep the above 5 recommendations close at hand to assist with their safe care. Also, be comfortable voicing your concern about prescribing safety with them so that they are also aware of the dangers scheduled drugs may carry. "If/when/then" is a form of "pre-suasion" that provides simple rules that tie goals to specific actions and has been used successfully to encourage behavior in many areas including medication adherence and drug abuse rehabilitation.
Arm/Group | Standard Letter | Comparator Letter
Number analyzed (Participants) | 269 | 241
Estimated average weekly MME dispensed
  52 weeks pre-letter | 157.70 [153.45 to 161.96] | 157.81 [153.85 to 161.76]
  4-52 weeks post-letter | 103.16 [100.34 to 105.98] | 89.96 [87.70 to 92.21]
Statistical Analysis 1: Comparison: Comparator Letter; Please note that 10% of means in the pre-intervention period were trimmed to remove outliers; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = -0.14, 95% CI 2-sided [-0.20 to -0.07], Standard Error of Mean 0.03 — This is the interaction coefficient for the difference-in-difference in average weekly MME pre-to-post letter between study arms. It was used to acquire the estimated average weekly MME post-letter in the Outcome Measure Data table

2. Secondary Outcome: Average Weekly Change in Valium Milligram Equivalents (VME) Dispensed.
Description: Difference in average weekly VME dispensed 52 weeks pre-letter to 4-52 (excludes 0-3 weeks for washout) post-letter. Measure of interest is the difference in the above measure between prescribers randomized to the standard letter and the comparator letter, referred to as the difference-in-difference (interaction coefficient).
Time Frame: 52 weeks pre-letter and 4-52 weeks post-letter (excludes 0-3 weeks for washout)
Population: Prescribers practicing in Los Angeles County with scheduled drug prescribing privileges who prescribed a benzodiazepine 52 weeks (1 year) prior to a patient death from a schedule II-IV overdose.
Measure: Mean (95% Confidence Interval); unit: Estimated average weekly VME dispensed
Arm/Group | Standard Letter | Comparator Letter
Number analyzed (Participants) | 277 | 251
Estimated average weekly VME dispensed
  52 weeks pre-intervention | 47.18 [45.90 to 48.46] | 43.09 [41.82 to 44.36]
  4-52 weeks post-intervention | 37.93 [36.93 to 38.94] | 31.77 [30.79 to 32.75]
Statistical Analysis 1: Comparison: Comparator Letter; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = -0.09, 95% CI 2-sided [-0.15 to -0.02], Standard Error of Mean 0.03 — This is the interaction coefficient for the difference-in-difference in average weekly MME pre-to-post letter between study arms. It was used to acquire the estimated average weekly VME post-letter in the Outcome Measure Data table

ADVERSE EVENTS:
Time Frame: 12 months following letter notification
Description: We hypothesize that there will be no difference in the proportion of prescribers in the intervention versus control group who make substantial (>20%) reductions in opioid prescribing in the post-intervention period.
Groups:
- Letter A Intervention: The intervention arm will involve letter A sent to prescribers in Los Angeles County.
  Letter A: The letter will be signed by the Chief Medical Examiner-Coroner and County Health Officer of Los Angeles County to notify prescribers of the death in their practice. The letter includes the decedent's name, date of birth and date of death, and outlines the annual number and types of prescription drug deaths seen by the medical examiner, discusses the value of and way to access the State's prescription drug monitoring program and includes five Centers for Disease Control and Prevention (CDC) guideline-recommended safe prescribing strategies: 1) Avoid co-prescribing of opioids with benzodiazepines, 2) prescribe minimal dose necessary for acute pain, 3) consider slow tapers with pauses to below 50 MME per day, 4) avoid prescriptions lasting greater than 3-months for pain, and 5) prescribe naloxone in conjunction with opioids for patients taking > 50 MME per day. The letter also states that CURES review is required by law as of October 2, 2018.
- Letter B Intervention: The intervention arm will involve letter B sent to prescribers in Los Angeles County.
  Letter B: This letter includes all the details in Letter A plus additional text involving an "if/when/then statement" along with an injunction to providers to share safety information with patients so that they identify as a "safe prescriber." Specifically, the additional text reads as follows: When your next patient presents with pain, keep the above 5 recommendations close at hand to assist with their safe care. Also, be comfortable voicing your concern about prescribing safety with them so that they are also aware of the dangers scheduled drugs may carry. "If/when/then" is a form of "pre-suasion" that provides simple rules that tie goals to specific actions and has been used successfully to encourage behavior in many areas including medication adherence and drug abuse rehabilitation.
Arm/Group | Letter A Intervention | Letter B Intervention
All-Cause Mortality (participants affected / at risk) | 0/269 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/269 | 0/241
Other Adverse Events (participants affected / at risk) | 0/269 | 0/241

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03856593/Prot_SAP_000.pdf